CLINICAL TRIAL: NCT01299337
Title: Acceleration and Relapse Prevention With Triiodothyronine (T3) as an Adjunct to Electroconvulsive Therapy (ECT)
Acronym: T3ECT
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Christopher Sola, D.O., Mayo Clinic
Other Study IDs: 07-004759
Record Dates: First submitted 2008-06-10; First posted 2011-02-18 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Triiodothyronine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Thyroid measures at time of sustained response will include free T3, free T4, and TSH. All draws will be done before ECT treatment. An additional free T3 will be obtained at the second visit that confirms sustained response. The mean free T3 will be used as the outcome measure. If a suppressed TSH is found, a TSH be repeated 1 week later. At the beginning of the study 30 mL of blood will be drawn and a portion of the collected blood sample will undergo DNA extraction. The extracted DNA will undergo genetic analysis. The remainder owill be immortalized and stored for future study. Blood will be drawn into 1 10-mL EDTA tube and 2 10-mL Heparin tubes . Samples will be stored at Mayo Clinic BAP Lab for subsequent DNA extraction, analysis, and storage.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- placebo: Subjects will be randomized either receiving T3 or placebo.
  Interventions: Drug: T3

INTERVENTIONS:
Drug: T3 — Given each day of ECT treatment 25 mg for the first 5 days increasing to 50 mg for the duration of treatment.
  Other Names: triiodythronine

SUMMARY:
The purpose of this study is:

* To evaluate liothyronine (Cytomel) as an accelerating agent (i.e. faster rate to clinical remission) to electroconvulsive therapy.
* To evaluate whether thyroid supplement acceleration can reduce the neurocognitive side effect of ECT treatment.
* To evaluate whether thyroid status at the time of remission is associated with subsequent relapse rate.
* To evaluate genetic polymorphisms in enzymes responsible for thyroid metabolism and the serotonin transporter promoter gene in depression (5-HTTLRP).

DETAILED DESCRIPTION:
This is a single-site, randomized, placebo-controlled trial of concurrent triiodothyronine (Cytomel® 25-50 mcg/d) to electroconvulsive therapy (ECT) in patients with a major depressive episode referred to ECT. Goals of this application are to: 1) evaluate whether thyroid status at time of sustained clinical response is associated with subsequent relapse rate, 2) evaluate triiodothyronine (Cytomel®) as an accelerating agent (i.e. faster rate to sustained clinical response) to electroconvulsive ECT treatment, and 3) evaluate whether thyroid acceleration can reduce the neurocognitive side effects of ECT. 4) To evaluate genetic polymorphisms in enzymes responsible for thyroid metabolism and the serotonin transporter promoter gene in depression (5-HTTLRP).

The primary outcome measure for this study, time to relapse, is defined as a Hamilton Depression Score (HAMD-24) ≥16 and an increase of ≥10 points from sustained response baseline. Secondary outcomes measures are time to sustained response, defined as a ≥60% reduction in the HAMD-24 score, and neurocognitive side effect burden as rated by the modified Mini Mental Status Examination at time of sustained clinical response.

Hypotheses:

1. Within a 6-month study period, mean serum free T3 at time of sustained clinical response will correlate with time to subsequent relapse [defined as a HAMD-24 score ≥16 with an increase of ≥10 points from baseline (sustained response)].
2. In comparison to placebo, triiodothyronine (Cytomel®, 25-50 mcg) will accelerate time to sustained clinical response [defined as a ≥60% reduction in the Hamilton Rating Scale for Depression, 24-item, (HAMD-24) score and a HAMD-24 total score ≤10 for 2 consecutive visits] in depressed patients referred to ECT.
3. In comparison to placebo, at time of sustained clinical response, there will be less ECT-related neurocognitive side effects, as rated by the modified Mini-Mental Status Examination (mMMSE), associated with triiodothyronine.
4. a. The 5-HTTLPR long allele (l) and (l)/(l) genotype will be associated with a faster treatment response.

   b. The DI-C785T allele will be associated with lower T3 levels at baseline and faster treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-64, male and female, any race/ethnicity
* Current diagnosis of major depression (unipolar)
* Currently Hospitalized at Mayo Clinic Physician recommendation for ECT treatment at Mayo Clinic
* Willing to return to Mayo Clinic for follow-up

Exclusion Criteria:

* Inability to speak English
* Inability or unwillingness to provide written informed consent
* Psychotic depression (SCID-confirmed)
* Court-ordered involuntary ECT
* Currently receiving maintenance ECT
* Unstable current medical condition
* A condition that would deem triiodothyronine treatment unsafe
* Diagnosis of primary thyroid disorder
* Lithium treatment within 6 weeks of randomization
* Currently taking levothyroxine (Synthroid®) or triiodothyronine (Cytomel®)
* Subclinical hypo- or hyperthyroidism
* History of atrial fibrillation or any cardiac arrhythmia except sinus bradycardia
* History of myocardial infarction within the past 12 months or unstable coronary artery disease
* Pregnancy
* History of Osteoporosis

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Consultants at the Department of Psychiatry and Psychology will evaluate patients with a diagnosis of depression (unipolar) for ECT. When a patient matches the study's diagnostic criteria, and does not meet any of the exclusion criteria, he/she will be asked to participate in the study.
  Patient will be contacted prior to first ECT Treatment by study personnel
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2008-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
To determine if people get better faster and stay better longer using T3 as adjunct to ECT. | Phase A and Phase B

CONTACTS AND LOCATIONS:
Overall Officials: Christopher L Sola, D.O., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Department of Psychiatry and Psychology, Rochester, Minnesota, United States